CLINICAL TRIAL: NCT06014125
Title: Tele-education in Patients With a Moderate Depressive Episode in Primary Care
Brief Title: Paramedical Tele-education on Moderate Depressive Episodes
Acronym: TE-DSP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: RC31/22/0262
Record Dates: First submitted 2023-08-22; First posted 2023-08-28 (Actual); Last update posted 2024-01-31 (Actual); Status verified 2024-01

CONDITIONS: Depression; Depression Moderate
Keywords: psychoeducation
MeSH Terms: conditions — Depression

STUDY DESIGN:
Intervention Model Description: Single-centered randomised controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- psychoeducation program group (Experimental): In addition to the usual treatment, the experimental group will receive a tele-education programme on depression in 5 individual remote sessions. During these sessions, the symptoms of the illness will be discussed, as well as health and diet measures, the destigmatisation of the illness, mobilisation of family and friends, the various treatments for depression and, finally, an assessment of what has been learned, which will be sent to the general practitioner with the patient's agreement.
  Interventions: Other: psychoeducative program
- control group (No Intervention): The control group will receive their usual care from their GP. An educational booklet on depression will be provided to patients at the start of the study.

INTERVENTIONS:
Other: psychoeducative program — The tele-education program consists of 5 sessions and is designed to adapt to changes in depressive symptoms over time. Each session will last an average of 60 minutes. They will be scheduled every week for 5 weeks.
  The first session is devoted to educational diagnosis, with identification of the patient's needs and any barriers to treatment.
  The second session will focus on personalised hygienic and dietary measures. A third session will focus on identifying the symptoms of depression, with a particular focus on suicidal ideation and the causes of depression. The role of family and friends will also be discussed.
  A fourth session will be devoted to providing clear information on antidepressants, with particular attention to the duration of treatment.
  The aim of the final session is to identify what has been learned and to clarify any questions before drawing up a joint summary of the work done, which will be sent to the patient's GP with his or her consent.
  Arms: psychoeducation program group

SUMMARY:
Considering that one out of five people may experience depression during the course of their life, and that compliance to anti-depression medication is often not optimal.

Psycho-educational interventions are recommended in international clinical practice guidelines for the management of depression. They are the first step in the treatment protocol.

Psychoeducation in the treatment of depressive episodes has been shown to be an effective intervention because it reduces depressive symptoms, the risk of relapse or recurrence and improves adherence to treatment.

In France, there are only one approved psycho-education programme, but it concerns a population of patients under psychiatric care.

No psycho-education programme has yet been carried out or evaluated in France on depressed patients followed up in primary care by their General Practitioner.

Recent changes in our healthcare practices, which have required adaptation to the pandemic context, have led to the development of the use of telemedicine.

This study aims to evaluate a new and 100% remote educational program adapted to patients ongoing moderate depression and focused on medication adherence, economic gain and patients and professional satisfaction.

DETAILED DESCRIPTION:
In addition to the usual standard care, recruited patients will benefit from either an individual tele-education programme or standard care following the randomisation.

The psycho-education programme is based on 3 dimensions: educational (nature of the information and how it should be delivered), psychological (revelation of the diagnosis and transmission of information in a personalised way), behavioural and cognitive (restoring the skills and mobilising the resources of the subject in their daily functioning and in their relationship with the disease (management of treatment and communication skills in particular).

A low number of sessions has been chosen, as it is more appropriate for this population, whose disorders are not severe and who do not require specialist care. The emphasis was placed on personalising the information, with one-to-one sessions.

The tele-education program consists of 5 sessions and is designed to adapt to changes in depressive symptoms over time. Each session will last an average of 60 minutes. They will be scheduled every week for 5 weeks.

The first session is devoted to educational diagnosis, with identification of the patient's needs and any barriers to treatment, in order to personalise the information to be provided about the programme.

The second session will focus on personalised hygienic and dietary measures. This will involve identifying sleep habits and leisure activities through behavioural analysis, and then identifying coping strategies with the patient in order to identify habits that can help combat depression.

A third session will focus on identifying the symptoms of depression, with a particular focus on suicidal ideation and the causes of depression. The role of family and friends will also be discussed.

A fourth session will be devoted to providing clear information on antidepressants, with particular attention to the duration of treatment.

The aim of the final session is to identify what has been learned and to clarify any questions before drawing up a joint summary of the work done, which will be sent to the patient's GP with his or her consent.

The liaison note is drawn up by the nurse with the patient for the general practitioner, focusing on: the patient's resources, in particular a personalised activity programme, and the patient's entourage, the areas of weakness identified and the risks identified of discontinuity in compliance.

Patients in the control group will receive standard care as usual. An educational booklet on depression, produced by the Institut National de Prévention et d'Education pour la Santé, will be sent to them by email after randomisation. It covers the symptoms, treatments and professionals to be consulted about depression. Patients will be able to consult this guide whenever they wish, without restriction, throughout the study.

Patients will usually be monitored by their General Practioner (GP), who may contact and refer them to the DSPP for psychiatric advice at any time during the study. The GP remains the referent for the patient's mental health care, with the support of the DSPP.

All participants in the study (control and experimental groups) may also be monitored by a psychologist, and will complete questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Presenting a depressive episode of moderate intensity according to the Diagnostic and Statistical Manual (DSM)-V
* With a prescription for an antidepressant started less than 2 months before inclusion in the trial.
* Whose state of health is compatible with follow-up by their GP (possibility of occasional advice from a psychiatrist).
* Have Internet access at home (computer) and are able to use the digital platform.

Exclusion Criteria:

* Patients who are unable to complete self-questionnaires (language barrier, etc.)
* Who have already undergone a psycho-education or therapeutic patient education programme regarding depression.
* Whose state of health requires follow-up by a psychiatrist

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2024-01-25 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
medication adherence | 6 months post inclusion
  The primary endpoint will be measured by the rate of maintenance on continuous antidepressant medication at 6 months after inclusion in the study.
  This maintenance rate will be measured using healthcare reimbursement data to reconstruct exposure to antidepressant medication at 6 months following inclusion in the study.

SECONDARY OUTCOMES:
Effectiveness of the tele-education | 3 months post inclusion
  Effectiveness of the tele-education programme compared with usual care on :
  1) Changes in feelings of self-efficacy using a scale of feelings of self-efficacy at inclusion and at 3 months: The investigators will use the General Self-Efficacy Scale (GSE). Each statement is scored from 1 to 4: "not at all true", "barely true", "moderately true" and "totally true". The scale contains ten items. This self-questionnaire will be completed by the patient via the digital platform at inclusion and 3 months post inclusion.
Effectiveness of the tele-education | 3 months post inclusion
  Effectiveness of the tele-education programme compared with usual care on :
  2) Changes in barriers to treatment using the Barriers to Care Evaluation (BACE) scale at inclusion and 3 months: The BACE-V3 scale is a self-administered questionnaire on barriers to access to care. It presents patients with possible barriers that may have prevented, delayed or discouraged them from seeking or pursuing professional care for a mental health problem. The help provided by a professional may be that of the GP, health staff (nurse, social worker, etc.), a psychiatrist, a counsellor, a psychologist or a psychotherapist. Patients are offered 4 response options for each of the 30 items, marked from 0 to 3: "not at all"; "a little"; "moderately"; "a lot".

OTHER OUTCOMES:
Evolution of depressive symptoms | 6 months post inclusion
  Evolution of PHQ-9 depressive symptoms:
  This will be carried out by comparing the differences in scores on the PHQ-9 scale at inclusion and at 6 months. The Patient Health Questionnaire-9 (PHQ-9) is a validated tool for assessing the severity of depressive disorder. The PHQ9 is a self-report screening tool. It contributes to the overall assessment of the patient and to monitoring his or her progress. The PHQ9 has been widely used and validated in primary care.
  It comprises nine items and respondents are asked to rate their experience of nine common symptoms of depression over the past two weeks.
  It is a 4-point rating scale where 0 indicates "not at all" and 3 "always".
  No depression: score from 0 to 4, Mild depression: score from 5 to 9, Moderate depression: score from 10 to 14, Moderately severe depression: score from 15 to 19 Severe depression: score from 20 to 27.

CONTACTS AND LOCATIONS:
Overall Officials: Marion LASSERRE, Principal Investigator — University Hospital, Toulouse
Locations (1):
- Chu Toulouse, Toulouse, Occitanie, France

IPD SHARING:
Plan to Share IPD: No